CLINICAL TRIAL: NCT03833531
Title: Prediction and Outcome Study in PTSD and (Cluster C) Personality Disorders
Brief Title: Effectiveness of PTSD-treatment Compared to Integrated PTSD-PD-treatment in Adult Patients With Comorbid PTSD and CPD
Acronym: PROSPER-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkin (Industry)
Collaborators: Sinai Centrum, Arkin, The Netherlands (Unknown); Amsterdam UMC, location VUmc (Other); Stichting Steunfonds Joodse Geestelijke Gezondheidszorg (SSF JGG) (Unknown); Ziekenhuis Amstelland (Other); Meander Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROSPER2018-C
Record Dates: First submitted 2019-01-24; First posted 2019-02-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Posttraumatic Stress Disorder (PTSD); Avoidant Personality Disorder; Dependent Personality Disorder; Obsessive Compulsive Personality Disorder
Keywords: PTSD; CPD; Imagination and rescripting therapy (ImRs); Schema-Focused Therapy (SFT); Integrated treatment; Prediction
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Personality Disorders; Dependent Personality Disorder; Compulsive Personality Disorder

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial comparing PTSD-treatment ImRs) to integrated PTSD-PD treatment (SFT-ImRS)in patients with PTSD and comorbid CPD.
  The PTSD treatment (ImRS) specifically address the troubling memories of the traumatic event and the personal meaning of the event and consist of 12 to 18 sessions in maximum 6 months. Integrated PTSD-PD treatment consist of a PTSD treatment (ImRS) interwoven in a PD treatment (SFT) that takes at least one group-session per week, for the duration of one year.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessments will be performed by allocation-blind assessors. Upon seeing a participant for an assessment, assessors are instructed to immediately state that participants are not allowed to discuss aspects of the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTSD-ImRS (Active Comparator): PTSD treatment
  Interventions: Behavioral: ImRS
- Integrated SFT-ImRS (Experimental): Integrated PTSD-PD treatment
  Interventions: Behavioral: ImRS; Behavioral: SFT

INTERVENTIONS:
Behavioral: ImRS — ImRs is a PTSD treatment that specifically addresses the troubling memories of the traumatic event and the personal meaning of the event and consist of 12 to 18 sessions in maximum 6 months.
Behavioral: SFT — SFT is a treatment for personality disorders that takes at least one group-session per week, for the duration of one year.
  Arms: Integrated SFT-ImRS

SUMMARY:
The goal of PROSPER-C is to study effectiveness of ImRs compared to integrated SFT-ImRs in treatment-seeking, adult patients with comorbid PTSD and Cluster C Personality Disorder (CPD).

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is highly comorbid with personality disorders (PD), mainly borderline (BPD) and cluster C personality disorders (CPD). It is not clear yet what treatment is most effective for those who suffer both PTSD and PD. There is growing preference in clinicians for evidence-based PTSD treatments, such as Eye Movement Desensitization and Reprocessing (EMDR) or Imagination and Rescripting (ImRs), because these treatments are relative short, and there is some evidence that comorbid PD symptoms might resolve as well. However, at least 30-44% PTSD patients do not sufficiently respond to PTSD treatments or are excluded because of suicidality or self-harm. PD treatments are more intensive than PTSD treatments, e.g. Dialectical Behavior Therapy (DBT) and Schema-Focused Therapy (SFT). There is some evidence that integrated PTSD-PD treatment is twice as effective than PD treatment alone, but integrated PTSD-PD treatment is not yet directly compared to PTSD treatment alone. This study will address this knowledge gap, including secondary outcome measures on functioning, quality of life and cost-effectiveness.

For patients with comorbid PTSD and CPD, ImRs-only will be compared to integrated SFT-ImRs (PROSPER-C).

Psychological (cognitive, affective, and relational) and neurobiological candidate predictors and mediators of treatment outcome will be investigated through a machine-learning paradigm, in order to develop a clinically useful and individual prediction instrument of treatment outcome. Example predictors and mediators are educational level , working memory, hyper- and hypo-arousal , therapeutic alliance and social support, resting state fMRI, an emotional face task fMRI , cortisol levels from hair samples and (epi)genetic markers.

For the neurobiological prediction, a subgroup of patients will undergo MRI scans, as will healthy controls as control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PTSD (309.81), and
* Diagnosed with a cluster C personality disorder (avoidant 301.82, dependent 301.6, and/or obsessive-compulsive PD 301.4), or at least resp. 3, 4, and/ or 3 criteria of these PDs.

To be eligible for the study, both patients and healthy controls (for the MRI scans) have to:

* Be aged between 18 and 65 years
* Give written informed consent
* Speak / understand Dutch sufficiently

Exclusion criteria:

* Current psychosis
* Comorbidity interfering with treatment or randomisation (severe outward aggression, antisocial PD, treatment interfering addiction or eating disorders, somatic problems)
* Primary diagnosis of paranoid, schizoid, schizotypal, narcissistic, histrionic or antisocial PD
* Mental retardation

Additional exclusion criteria for the MRI substudy are:

* Pregnancy
* Metal implants (such as pacemakers, etc.);
* Somatic disorders interfering with brain functioning
* Claustrophobia
* High dose use of benzodiazepines

For the healthy controls, current psychiatric diagnosis is an additional exclusion criterion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
CAPS-5 (Clinician Administered PTSD Scale) | 12 months
  The CAPS-5 is a structured diagnostic interview to assess the frequency and severity of DSM-5 PTSD symptoms. The interview consists of 30 items, with higher scores indicating more severe symptomatology. CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms. Similarly, CAPS-5 symptom cluster severity scores are calculated by summing the individual item severity scores for symptoms corresponding to a given DSM-5 cluster: Criterion B (items 1-5); Criterion C (items 6-7); Criterion D (items 8-14); and, Criterion E (items 15-20). A symptom cluster score may also be calculated for dissociation by summing items 19 and 20. To meet the criteria for PTSD diagnoses, at least one Criterion B and one Criterion C symptom, and two criterion D and E symptoms are required. Furthermore, Criterion F and G should be met.

SECONDARY OUTCOMES:
SCID-5-PD (Structured Interview for DSM-5 Personality Disorders) | 12 months
  The SCID-5-PD is a semi-structured interview to assess the presence and severity of the DSM-5 personality disorders. Diagnoses are made either categorically (present or absent) or dimensionally (summing the ratings for each symptom. The symptoms are rated 0, 1 or 2).
PCL-5 (PTSD Checklist for DSM-5) | 12 months
  The PCL-5 is a self-reported PTSD symptom scale. It consists of 20 items, scored 0 ("not at all") to 4 ("Extremely"). This is summed for total self-reported PTSD-severity, range 0 (no self-reported PTSD-symptoms in the past month) to 80 (extreme self-reported PTSD-symptoms in the past month). There are subscales for the different PTSD symptom clusters; cluster B (question 1-5), C (6-7); D (8-14) and E (15-20).
OQ-45 (Outcome Questionnaire-45) | 12 months
  The OQ-45 is a self-report questionnaire that measures general functioning and physical complaints in the past week. It consists of 45 items; 25 items on psychiatric symptoms and 20 on interpersonal, occupational and social functioning. These are rated from 0 ("Never") to 4 ("Almost always"). Some items need to be reversed in scoring. There are four subscales: Symptomatic Distress (25 items); Interpersonal Relationships (11 items) and Social Role (9 items). A higher score indicates worse functioning.
BDI (Beck depression inventory) | 12 months
  The BDI is a 21-item self-report questionnaire assessing the severity of depression. Each item consists of four statements indicating different levels of severity of a particular symptom experienced over the past week, ranging from low (0) to high (3) severity. Scores for all 21 items are summed to yield a single depression, with a maximum depression score of 63.
AUDIT (Alcohol Use Disorders Identification Test) | 12 months
  The AUDIT is a self-report questionnaire, with 10 items about alcohol use. These range from 0 ("Never") to 4 ("Daily"). The items are summed to create a total score from 0 (no alcohol risk) to 40 (maximum alcohol risk). The first three questions are about alcohol consumption, question 4-6 about alcohol dependency and question 7-10 about alcohol related problems.
SCID-5-S (Structured Clinical Interview for DSM-5 Disorders - syndrome disorders) | 12 months
  The SCID-5-S is a clinician administered semistructured clinical interview to assess DSM-5 disorders (but not personality disorders). It consists of in total 14 modules, comparable to the DSM-5. Patients are assessed on the disorder, resulting in a score of absent/present for each disorder. In this study, we use the modules current depressive episode, current manic episode, current persistent depressive disorder, delusions & hallucinations, alcohol abuse, substance abuse, panic disorder, agoraphobia, specific phobia, generalized anxiety disorder, obsessive-compulsive disorder, current anorexia, bulimia and binge eating disorder.
WHODAS 2.0 (World Health Organization Disability Assessment Schedule) | 12 months
  WHODAS 2.0 is a 36-item self-report questionnaire assessing the daily function of activity and participation within the 30 previous days, including the following six domains: Cognition, Mobility, Self-care, Getting along, Life activities and Participation. The responses on each item range from no difficulty (1) to extreme difficulty (5). Responses to the six dimensions are weighted and summed to create a total score between 0 (no disability) and 100 (complete disability).
EQ-5D-5L (EuroQOL - 5 Dimensions - 5 Levels) | 12 months
  The EQ-5D-5L measures health-related quality of life and consists of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The answer to each item results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state, with higher numbers indicating more severe problems.
Tic-P (Trimbos/iMTA questionnaire for costs associated with psychiatric illness) | 12 months
  TiC-P is a self-report questionnaire assessing direct medical costs and productivity costs due to absence from work or reduced efficiency during work in patients with a mental disorder. The first part of the TiC-P includes 14 structured yes or no questions on the use of medical resources, each followed by a question on the volume of medical consumption. The second part includes five items on work absence, reduced efficiency at work and related productivity losses.
NSSI (Non-Suicidal Self-Injury) | 12 months
  The NSSI screener consists of 7 multiple-choice items assessing non-suicidal self-injury. In case of an affirmative responses to the item 'Have you ever done any of the following with the purpose of intentionally hurting yourself?' engagement in NSSI is determined.
PAI-BOR (Personality Assessment Inventory- Borderline features scale) | 12 months
  The Personality Assessment Inventory-Borderline Features (PAI-BOR) Scale is a self-report measure assessing the presence and severity of BPD. The BAI-BOR consists of four subscales of six items each, reflecting four main characteristics of BPD: affective instability, negative relationships, identity problems and self-harm. Each items is rated on a four-point scale, ranging from false (0) to very true (3). A total PAI-BOR score of 38 or more indicates the presence of significant BPD features, whereas a score of 60 or more indicates typical borderline personality functioning.
YSQ-75 (Young Schema Questionnaire - 75 Items) | 12 months
  The YSQ-75 is a 75-item self-report questionnaire assesses 15 schemas: temporally stable, personal and interpersonal patterns of beliefs, feelings, sensations and thoughts. Items are rated on a 6-point scale ranging from 1 = Completely untrue of me to 6 = Describes me perfectly. There is evidence for adequate validity and reliability values. Although sparse, evidence suggests that dysfunctional schema reduction accompanies personality disorder symptom reduction after ST.
SMI-118 (Schema Mode Inventory - 118 Items) | 12 months
  The SMI-118 is a 118-item self-report questionnaire assessing 14 schema modes, defined as "those schemas or schema operations - adaptive or maladaptive - that are currently active for an individual". Each item is rated on a 6-point scale ranging from 1 (never) to 6 (always). Adequate psychometric properties have been reported. Although sparse, evidence suggests that dysfunctional schema mode reduction accompanies symptom reduction after ST. Similar to dysfunctional schema reduction, evidence suggests that dysfunctional schema mode reduction accompanies personality disorder symptom reduction after ST.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Thomaes, MD/PhD, Principal Investigator — Sinai Centre
Locations (1):
- Sinai Centrum, Amstelveen, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
There is no concrete plan for sharing yet, possibly neurobiological and (epi)genetic data will be shared in a later stage. Patients are asked to sign consent forms for future data sharing.

REFERENCES:
- [Background] Bradley R, Greene J, Russ E, Dutra L, Westen D. A multidimensional meta-analysis of psychotherapy for PTSD. Am J Psychiatry. 2005 Feb;162(2):214-27. doi: 10.1176/appi.ajp.162.2.214. PMID 15677582
- [Background] Harned MS, Korslund KE, Linehan MM. A pilot randomized controlled trial of Dialectical Behavior Therapy with and without the Dialectical Behavior Therapy Prolonged Exposure protocol for suicidal and self-injuring women with borderline personality disorder and PTSD. Behav Res Ther. 2014 Apr;55:7-17. doi: 10.1016/j.brat.2014.01.008. Epub 2014 Feb 11. PMID 24562087
- [Background] Ehlers A, Clark DM, Hackmann A, McManus F, Fennell M. Cognitive therapy for post-traumatic stress disorder: development and evaluation. Behav Res Ther. 2005 Apr;43(4):413-31. doi: 10.1016/j.brat.2004.03.006. PMID 15701354
- [Background] Lanius RA, Vermetten E, Loewenstein RJ, Brand B, Schmahl C, Bremner JD, Spiegel D. Emotion modulation in PTSD: Clinical and neurobiological evidence for a dissociative subtype. Am J Psychiatry. 2010 Jun;167(6):640-7. doi: 10.1176/appi.ajp.2009.09081168. Epub 2010 Apr 1. PMID 20360318
- [Background] Nijdam MJ, de Vries GJ, Gersons BP, Olff M. Response to psychotherapy for posttraumatic stress disorder: the role of pretreatment verbal memory performance. J Clin Psychiatry. 2015 Aug;76(8):e1023-8. doi: 10.4088/JCP.14m09438. PMID 26335088
- [Background] van Rooij SJ, Kennis M, Vink M, Geuze E. Predicting Treatment Outcome in PTSD: A Longitudinal Functional MRI Study on Trauma-Unrelated Emotional Processing. Neuropsychopharmacology. 2016 Mar;41(4):1156-65. doi: 10.1038/npp.2015.257. Epub 2015 Aug 20. PMID 26289143
- [Background] Cloitre M, Stovall-McClough KC, Miranda R, Chemtob CM. Therapeutic alliance, negative mood regulation, and treatment outcome in child abuse-related posttraumatic stress disorder. J Consult Clin Psychol. 2004 Jun;72(3):411-6. doi: 10.1037/0022-006X.72.3.411. PMID 15279525
- [Background] Bryant RA, Felmingham K, Kemp A, Das P, Hughes G, Peduto A, Williams L. Amygdala and ventral anterior cingulate activation predicts treatment response to cognitive behaviour therapy for post-traumatic stress disorder. Psychol Med. 2008 Apr;38(4):555-61. doi: 10.1017/S0033291707002231. Epub 2007 Nov 16. PMID 18005496
- [Background] Brewin CR, Andrews B, Valentine JD. Meta-analysis of risk factors for posttraumatic stress disorder in trauma-exposed adults. J Consult Clin Psychol. 2000 Oct;68(5):748-66. doi: 10.1037//0022-006x.68.5.748. PMID 11068961
- [Background] Bisson J, Andrew M. Psychological treatment of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2007 Jul 18;(3):CD003388. doi: 10.1002/14651858.CD003388.pub3. PMID 17636720
- [Background] Bisson JI, Roberts NP, Andrew M, Cooper R, Lewis C. Psychological therapies for chronic post-traumatic stress disorder (PTSD) in adults. Cochrane Database Syst Rev. 2013 Dec 13;2013(12):CD003388. doi: 10.1002/14651858.CD003388.pub4. PMID 24338345
- [Background] Clarke SB, Rizvi SL, Resick PA. Borderline personality characteristics and treatment outcome in cognitive-behavioral treatments for PTSD in female rape victims. Behav Ther. 2008 Mar;39(1):72-8. doi: 10.1016/j.beth.2007.05.002. Epub 2007 Oct 22. PMID 18328872
- [Background] Frias A, Palma C. Comorbidity between post-traumatic stress disorder and borderline personality disorder: a review. Psychopathology. 2015;48(1):1-10. doi: 10.1159/000363145. Epub 2014 Sep 9. PMID 25227722
- [Background] Feeny NC, Zoellner LA, Foa EB. Treatment outcome for chronic PTSD among female assault victims with borderline personality characteristics: a preliminary examination. J Pers Disord. 2002 Feb;16(1):30-40. doi: 10.1521/pedi.16.1.30.22555. PMID 11881159
- [Background] Hembree EA, Cahill SP, Foa EB. Impact of personality disorders on treatment outcome for female assault survivors with chronic posttraumatic stress disorder. J Pers Disord. 2004 Feb;18(1):117-27. doi: 10.1521/pedi.18.1.117.32767. PMID 15061348
- [Background] Stoffers JM, Vollm BA, Rucker G, Timmer A, Huband N, Lieb K. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD005652. doi: 10.1002/14651858.CD005652.pub2. PMID 22895952
- [Background] Kredlow MA, Szuhany KL, Lo S, Xie H, Gottlieb JD, Rosenberg SD, Mueser KT. Cognitive behavioral therapy for posttraumatic stress disorder in individuals with severe mental illness and borderline personality disorder. Psychiatry Res. 2017 Mar;249:86-93. doi: 10.1016/j.psychres.2016.12.045. Epub 2017 Jan 4. PMID 28086181
- [Background] Roberts BW, Luo J, Briley DA, Chow PI, Su R, Hill PL. A systematic review of personality trait change through intervention. Psychol Bull. 2017 Feb;143(2):117-141. doi: 10.1037/bul0000088. Epub 2017 Jan 5. PMID 28054797
- [Background] Raabe S, Ehring T, Marquenie L, Olff M, Kindt M. Imagery Rescripting as stand-alone treatment for posttraumatic stress disorder related to childhood abuse. J Behav Ther Exp Psychiatry. 2015 Sep;48:170-6. doi: 10.1016/j.jbtep.2015.03.013. Epub 2015 Apr 4. PMID 25898289
- [Background] Arntz A, Tiesema M, Kindt M. Treatment of PTSD: a comparison of imaginal exposure with and without imagery rescripting. J Behav Ther Exp Psychiatry. 2007 Dec;38(4):345-70. doi: 10.1016/j.jbtep.2007.10.006. Epub 2007 Oct 26. PMID 18005935
- [Background] Farrell JM, Shaw IA, Webber MA. A schema-focused approach to group psychotherapy for outpatients with borderline personality disorder: a randomized controlled trial. J Behav Ther Exp Psychiatry. 2009 Jun;40(2):317-28. doi: 10.1016/j.jbtep.2009.01.002. Epub 2009 Jan 14. PMID 19176222
- [Derived] van den End A, Beekman ATF, Dekker J, Aarts I, Snoek A, Blankers M, Vriend C, van den Heuvel OA, Thomaes K. Trauma-focused and personality disorder treatment for posttraumatic stress disorder and comorbid cluster C personality disorder: a randomized clinical trial. Eur J Psychotraumatol. 2024;15(1):2382652. doi: 10.1080/20008066.2024.2382652. Epub 2024 Aug 1. PMID 39087734
- [Derived] Aarts I, Vriend C, Snoek A, van den End A, Blankers M, Beekman ATF, Dekker J, van den Heuvel OA, Thomaes K. Neural correlates of treatment effect and prediction of treatment outcome in patients with PTSD and comorbid personality disorder: study design. Borderline Personal Disord Emot Dysregul. 2021 May 5;8(1):13. doi: 10.1186/s40479-021-00156-8. PMID 33947471
- [Derived] van den End A, Dekker J, Beekman ATF, Aarts I, Snoek A, Blankers M, Vriend C, van den Heuvel OA, Thomaes K. Clinical Efficacy and Cost-Effectiveness of Imagery Rescripting Only Compared to Imagery Rescripting and Schema Therapy in Adult Patients With PTSD and Comorbid Cluster C Personality Disorder: Study Design of a Randomized Controlled Trial. Front Psychiatry. 2021 Mar 19;12:633614. doi: 10.3389/fpsyt.2021.633614. eCollection 2021. PMID 33868050

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT03833531/Prot_SAP_001.pdf